CLINICAL TRIAL: NCT06706401
Title: A Multicenter, Randomised 2*2 Factorial Design Comparing Standard to Reduced-target Volume Radiotherapy With or Without All-trans Retinoic Acid (ATRA) in Patients With Lateralised Oropharyngeal, Laryngeal and Hypopharyngeal Squamous Cell Carcinoma.
Brief Title: Lymphocyte-Sparing And Radio-Immunotherapy in Head and Neck Carcinoma
Acronym: Lysari
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Centre Leon Berard (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: ET 22-156
Record Dates: First submitted 2024-11-19; First posted 2024-11-26 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Oropharynx Cancer; Larynx Cancer; Hypopharynx Cancer; Primary Head and Neck Tumor
Keywords: Localised squamous cell carcinoma of head and neck; Previously untreated; Standard radiotherapy; Tailored radiotherapy; Vesanoid
MeSH Terms: conditions — Oropharyngeal Neoplasms; Laryngeal Neoplasms; Hypopharyngeal Neoplasms; Head and Neck Neoplasms | interventions — Tretinoin; Cisplatin; Cetuximab

STUDY DESIGN:
Intervention Model Description: This trial is a 2*2 factorial design, multicentric, randomised, Phase III study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Standard radiotherapy (Active Comparator): Patient will receive 6 to 8 weeks of standard (chemo)radiotherapy then will be followed until document progression disease, death, withdrawal of consent or end of trial (whichever occurs first).
  In addition of radiotherapy, patient will receive cisplatin or cetuximab (standard of care treatments).
  Interventions: Radiation: Standard radiotherapy; Drug: Cisplatin; Drug: Cetuximab
- Tailored radiotherapy and ATRA (Vesanoid) (Experimental): ATRA will be administered per os 1 week before the start of (chemo)radiotherapy (daily administration for 3 days). Then, patient will receive 6 to 8 weeks of tailored (chemo)radiotherapy. In addition of radiotherapy, patient will receive cisplatin or cetuximab (standard of care treatments). Subsequently, ATRA will be administered per os for 3 days every 3 weeks for a total of 4 courses starting 2 to 3 weeks after the end of (chemo)radiotherapy. Finally, the patient will be followed until document progression disease, death, withdrawal of consent or end of trial (whichever occurs first).
  Interventions: Drug: Vesanoid; Radiation: Tailored radiotherapy; Drug: Cisplatin; Drug: Cetuximab
- Standard radiotherapy and ATRA (Vesanoid) (Experimental): ATRA will be administered per os 1 week before the start of (chemo)radiotherapy (daily administration for 3 days). In addition of radiotherapy, patient will receive cisplatin or cetuximab (standard of care treatments).Then, patient will receive 6 to 8 weeks of standard (chemo)radiotherapy. Subsequently, ATRA will be administered per os for 3 days every 3 weeks for a total of 4 courses starting 2 to 3 weeks after the end of (chemo)radiotherapy. Finally, the patient will be followed until document progression disease, death, withdrawal of consent or end of trial (whichever occurs first).
  Interventions: Drug: Vesanoid; Radiation: Standard radiotherapy; Drug: Cisplatin; Drug: Cetuximab
- Tailored radiotherapy (Experimental): Patient will receive 6 to 8 weeks of tailored (chemo)radiotherapy then will be followed until document progression disease, death, withdrawal of consent or end of trial (whichever occurs first).
  In addition of radiotherapy, patient will receive cisplatin or cetuximab (standard of care treatments).
  Interventions: Radiation: Tailored radiotherapy; Drug: Cisplatin; Drug: Cetuximab

INTERVENTIONS:
Drug: Vesanoid — Before (chemo)radiotherapy: D1 to D3: 150mg/m2/day, 1 week before radiotherapy. Post (chemo)radiotherapy: D1 to D3: 150mg/m2/day every 3 weeks for up to 4 cycles post (chemo)radiotherapy
  Other Names: ATRA
  Arms: Standard radiotherapy and ATRA (Vesanoid); Tailored radiotherapy and ATRA (Vesanoid)
Radiation: Standard radiotherapy — 70 Gy in 35 fractions of 2 Gy over 6 (6 fractions per week) or hyperfractionated RT with a median therapeutic dose of 80.5 Gy delivered in 70 fractions of 1.15 Gy over 7 weeks.
  Arms: Standard radiotherapy; Standard radiotherapy and ATRA (Vesanoid)
Radiation: Tailored radiotherapy — 70 Gy in 35 fractions of 2 Gy over 6 weeks (6 fractions per week) or hyperfractionated RT with a median therapeutic dose of 80.5 Gy delivered in 70 fractions of 1.15 Gy over 7 weeks.
  Arms: Tailored radiotherapy; Tailored radiotherapy and ATRA (Vesanoid)
Drug: Cisplatin — Cisplatin is recommended for the following patients : Stage T1-T2/N2a-N2b and T3/N0-N1-N2a-N2b. concomitant chemotherapy is standard of care treatments and should be administered as per standard practice.
  Chemotherapy will include one of the two cisplatin regimens specified in this protocol at the discretion of the participating centers. The centers must however treat all their recruited patients with one of the two regimens chosen before site activation. Chemotherapy should start the first day of radiotherapy. Cisplatin should be infused before radiation therapy delivery.
  The 2 options are:
  • Cisplatin 100 mg/m² i.v. on day 1 and 22 of radiotherapy (when 70 Gy are delivered in 6 weeks) or on day 1, 22 and 43 (when 70 Gy are delivered in 7 weeks).
  or
  • Cisplatin 40 mg/m² i.v. on day 1, 8, 15, 22, 29, 35 of radiotherapy (when 70 Gy are delivered in 6 weeks) or on day 1, 8, 15, 22, 29, 35, 42 of radiotherapy (when 70 Gy are delivered in 7 weeks).
Drug: Cetuximab — Cetuximab is recommended for the following patients : Stage T1-T2/N2a-N2b and T3/N0-N1-N2a-N2b. concomitant Cetuximab is standard of care treatments and should be administered as per standard practice.
  Cetuximab therapy will be started with an intravenous loading dose of 400 mg/m2 one week before start of RT followed by six (radiotherapy over 6 weeks) or seven (radiotherapy over 7 weeks) weekly doses of 250 mg/m2.

SUMMARY:
The aim of this study is to investigate the effect of ATRA (Vesanoid) and the effect of tailored radiotherapy in patients with squamous cell carcinoma of the oropharynx, larynx or hypopharynx.

DETAILED DESCRIPTION:
Following validation of eligibility criteria, patients will be randomised (1:1:1:1) to receive:

* Arm A: Standard radiotherapy then follow-up
* Arm B: Tailored radiotherapy and ATRA (Vesanoid)
* Arm C: Standard radiotherapy and ATRA (Vesanoid)
* Arm D: Tailored radiotherapy then follow-up

This randomised phase III clinical trial will provide the clinical proof-of-concept that unilateral irradiation for lateralized tumors and the addition of ATRA (Vesanoid) to radiotherapy in HNSCC prevents severe lymphopenia and immunosenescence and therefore, may foster a radiation-induced anticancer immune response sufficient to increase event-free survival at 2 years.

ELIGIBILITY:
Inclusion criteria :

I1. Male or female patients aged ≥ 18 years old at time of inform consent signature.

I2. Patients with primary head and neck tumour up to, but not crossing the midline, previously untreated with histologically-confirmed squamous cell carcinoma of:

* the oropharynx p16-, larynx or hypopharynx : T1/N2a-N2b, T2/N0-N2b, T3/N0-N2b (UICC 8th Ed.), or
* the oropharynx p16+ : T1/N1 (multiple nodes), T2-T3/N0-N1 (UICC 8th Ed.).

I3. Patients with lymph node staging assessed by an FDG-PET/CT with no contralateral nodal uptake.

I4. Patients amenable to treatment with RT or concomitant chemo-radiotherapy as decided by the treating physician as a function of tumor stage, tumor location, performance of the patients.

I5. Eastern Cooperative Oncology Group (ECOG) Performance Status 0 or 1.

I6. Adequate hematologic and end-organ function, defined by the following laboratory test results obtained within 7 days prior to randomisation :

Hematological (without transfusion within 2 weeks) :

* Neutrophils count > 1.5 × 109 /L
* Platelets count > 75 × 109 /L
* WBC≥ 3.0 × 109 /L

Hepatic function :

* Total Bilirubin < 1.5 × ULN (except for Gilbert's syndrome which will allow bilirubin ≤ 3 ULN).
* Alanine aminotransferase (ALT) ≤ 2.5 × ULN.
* Aspartate aminotransferase (AST) ≤ 2.5 × ULN.
* Albumin >3.0g/dL

Renal function :

* Serum creatinine < 1.5 ×ULN.

I7. QTcF ≤450ms for men and 470ms for women, from 3 electrocardiograms on screening ECG, within 7 days prior randomisation.

I8. Women patients of child-bearing potential are eligible, provided they have a negative serum or urine pregnancy test within 7 days prior randomisation, and agrees to use adequate contraception for up to 1 month after the end of study treatments.

I9. Fertile men must agree to use an effective method of contraception during the study and for up to 1 month after the end of study treatments.

I10. Patient should understand, sign, and date the written voluntary informed consent form prior to any protocol-specific procedures performed and should be able and willing to comply with study visits and procedures as per protocol.

I11. Patients must be covered by a medical insurance in country where applicable.

Exclusion criteria :

E1. Patient with primary tumor crossing the midline or patients with bilateral primary tumors.

E2. Patients with T1-N0 (p16-), T1-N1 (p16-), T1-N0 (p16+), T4 (p16- and p16+), bilateral lymph nodes or nodal disease more than 6 cm (p16- and p16+).

E3. Patients with unknown primary tumor size as per TNM i.e. T0-N1 to T0-N3, p16- or p16+.

E4. Patients with contralateral FDG-PET/CT nodal uptake.

E5. Patient with any previous anti-cancer therapy for HNSCC (all prior treatment are forbidden: chemotherapy, radiotherapy, targeted therapy, immunotherapy or any other therapy approved or experimental).

E6. Patient with malignancies other than HNSCC within 3 years prior to randomisation with the exception of adequately treated carcinoma in situ of the cervix, basal or squamous cell skin cancer, localised prostate cancer treated surgically with curative intent.

E7. Patient with ongoing or anticipation of need for systemic immunosuppressive medication (including, but not limited to, glucocorticoids, corticosteroids, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-TNF-alpha agents); with the exceptions of intranasal, inhaled or topical corticosteroids or systemic corticosteroids at physiological doses, which are not to exceed 10 mg/day of prednisone, or an equivalent corticosteroid.

E8. Patient with ongoing or anticipation of need for systemic immunostimulatory agents (including, but not limited to, interferons and IL-2).

E9. Patient with concurrent treatment with any other anti-cancer treatment, approved or investigational agent or participation in another clinical trial with therapeutic intent.

E10. Patient with infectious diseases :

* Severe infection within 4 weeks prior to randomisation, including, but not limited to, hospitalization for complications of infection, bacteremia, or severe pneumonia,
* Active hepatitis B (chronic or acute; defined as having a positive hepatitis B surface antigen [HBsAg] test at screening),
* Active hepatitis C. Patients positive for hepatitis C virus (HCV) antibody are eligible only if PCR is negative for HCV RNA at screening,
* HIV infection,
* Active tuberculosis.

E11.Patient with any psychological, cognitive, familial, sociological or geographical condition potentially hampering compliance with the study protocol, completion of patient reported measures and follow-up schedule; those conditions should be discussed with the patient before registration in the trial.

E12. Patient with known hypersensitivity to tretinoin, other retinoids, soya, peanut or to any of the excipients of vesanoid.

E13. Patient with known malabsorption syndrome and/or unable to swallow oral medication.

E14.Patient with ongoing or expected need for concomitant treatment with vitamin A, tetracyclines, other retinoids, anti-fibrinolytic agent, and strong inducers or inhibitors of CYP3A4.

E15.Pregnant or lactating woman.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 460 (Estimated)
Dates: Start 2025-02-20 (Actual); Primary Completion 2029-01 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
Event Free Survival (EFS) | At 6, 9, 15, 21 and 27 months from randomisation then annually assessed up to 2 years
  Event free survival (EFS) is defined as the time from randomisation to apparition of a documented relapse either local or regional or distant according to clinical or radiological assessment, or persistent residual disease including pathologically positive neck node, or death due to any cause.

SECONDARY OUTCOMES:
Local relapse Free Survival | At 6, 9, 15, 21 and 27 months from randomisation then annually assessed up to 2 years
  Local relapse Free Survival (lrFS, at site of primary tumor) is defined as the delay from randomisation to first local relapse (i.e. primary site) or death. Patients without documented event will be censured at the last adequate visit or tumor evaluation.
Regional relapse Free survival | At 6, 9, 15, 21 and 27 months from randomisation then annually assessed up to 2 years
  Regional relapse Free survival (rrFS, in the neck) is defined as the delay from randomisation to first regional relapse (i.e. neck) or death.
Metastasis Free Survival | At 6, 9, 15, 21 and 27 months from randomisation then annually assessed up to 2 years
  Metastasis Free Survival (mFS) is the time between randomisation and apparition of first metastasis (date of metastatic diagnosis). Patients without documented event will be censured at the last tumour evaluation.
Rate of pathologically positive lymph nodes | At 4 months from the completion of (chemo)-radiotherapy
  Rate of pathologically positive lymph nodes at neck node dissection performed at 4 months after the completion of (chemo)-radiotherapy for those patients benefiting from a neck node dissection
Event Free Survival (EFS) | At 4 months from the completion of (chemo)-radiotherapy
  Event Free Survival (EFS) considering that pathologically positive neck node within 4 months post-randomisation will not be an event.
Overall survival | Until up to 2 years follow-up of the last patient enrolled
  Overall survival defined as the time from randomisation to death due to any cause. Patient without documented death at the time of analysis will be censored at the date of last known contact.
Adverse events | From the date of first intake of study drug until 27 months after the randomisation of the last randomised patient
  Incidence of any adverse events graded according to NCI-CTCAE V5.0
Patient quality of life (EORTC QLQ-C30) | At randomisation, at 6, 9, 15, 21 and 27 months after randomisation and30 days after the last study treatments administration
  To assess the impact of the proposed combinations on patient' quality of life in the target population (EORTC QLQ-C30)
Patient quality of life (EQ5-DL) | At randomisation, at 6, 9, 15, 21 and 27 months after randomisation and30 days after the last study treatments administration
  To assess the impact of the proposed combinations on patient' quality of life in the target population (EQ5-DL)
Patient quality of life (EORTC QLQ-H&N43) | At randomisation, at 6, 9, 15, 21 and 27 months after randomisation and30 days after the last study treatments administration
  To assess the impact of the proposed combinations on patient' quality of life in the target population (EORTC QLQ-H&N43)
Health economic analysis | From the first patient enrolled to 2 years after treatment discontinuation of the last patient enrolled
  To perform an economic analysis of the use of a tailored-RT with or without ATRA (Vesanoid). A cost-effectiveness methodology will be implemented, which involves computing costs and efficacy for each of the four treatment arms.
Immunomonitoring | Cycle 1 Day 1 pre-dose of Vesanoid, Day 1 of radiotherapy and end of radiotherapy (8 to 10 weeks after randomisation)
  To study the impact of treatment on lymphocytes number and function, including by assessing immunosenescence induction and to study blood biomarkers predictive of response/toxicity following treatment

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Grégoire, PhD, Principal Investigator — Centre Leon Berard
Locations (7):
- France (7):
  - Institut de Cancérologie de l'Ouest - Paul Papin, Angers
  - Centre Oscar Lambret, Lille
  - Centre Léon Bérard, Lyon
  - Centre Antoine Lacassagne, Nice
  - AP-HP - Hôpital Tenon, Paris
  - Institut de Cancérologie de Lorraine, Vandœuvre-lès-Nancy
  - Institut Gustave Roussy, Villejuif